CLINICAL TRIAL: NCT01038375
Title: Tailored Interventions to Improve Hypertension Management After Stroke or TIA
Brief Title: Tailored Interventions to Improve Hypertension Management After Stroke or Transient Ischemic Attack (TIA)
Acronym: TIMSII
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, Gail MacKenzie, Clinical Nurse Specialist, Stroke Prevention Clinic, Hamilton Health Sciences, General Site, McMaster University
Organization: McMaster University (Other)
Other Study IDs: OSN0912-000106
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Blood Pressure
Keywords: hypertension; stroke; adherence
MeSH Terms: conditions — Hypertension; Stroke | interventions — Motivational Interviewing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Adherence counseling
  Interventions: Behavioral: lifestyle counseling, home blood pressure monitoring
- Usual care
  Interventions: Behavioral: lifestyle counseling, home blood pressure monitoring

INTERVENTIONS:
Behavioral: lifestyle counseling, home blood pressure monitoring — monthly telephone counseling over 6 months for intervention group no health provider initiated contact for control group
  Other Names: motivational interviewing

SUMMARY:
The purpose of this study is to determine the effectiveness of interventions to improve adherence to medication and healthier lifestyle choices on blood pressure over a 6 month period in a group of people at high risk for recurrent stroke events. The participants have already had a stroke or TIA, and have uncontrolled blood pressure, as well as problems with memory and problem-solving, or miss taking medications, or who do not believe in the effectiveness of their medications. Interventions focus on motivational interviewing, adherence counseling with memory cuing, and self-monitoring of blood pressure.

DETAILED DESCRIPTION:
* randomized, controlled trial at 4 sites
* measurement of blood pressure, missed pills, self-efficacy rating at baseline and 6 months
* contacting family pharmacists to evaluate prescription renewal patterns at baseline and 6 months

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of stroke or TIA
* hypertension
* Montreal Cognitive Assessment score less than 26
* self report of missed pills
* self-efficacy rating less than 100%

Exclusion Criteria:

* inability to give informed consent
* 18 years of age or younger

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clients recruited from Stroke Prevention Clinics in Ontario with diagnosis of Stroke or TIA, Hypertension, and cognitive deficits as indicated by MoCA score < 26, self-efficacy rating < 100%, and self-report of missed pills; English speaking; able to give informed consent; older than 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
blood pressure | 6 months from baseline testing

SECONDARY OUTCOMES:
self-efficacy rating | 6 months from baseline

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Royal Victoria Hospital, Barrie, Ontario
  - Hamilton General Hospital, 237 Barton St East, Hamilton, Ontario
  - Lakeridge Health Centre, Oshawa, Ontario